CLINICAL TRIAL: NCT04299373
Title: Effects of Metabolic Surgery on Alcohol Pharmacokinetics
Brief Title: Surgical Weight Loss and Alcohol Perception
Acronym: SWAP
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: In an effort to seek a more suitable method to measure alcohol clearance.
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Bruce Bartholow, Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016390
Record Dates: First submitted 2020-02-12; First posted 2020-03-06 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Bariatric Surgery Candidate
Keywords: metabolic surgery; alcohol; bariatric surgery
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two routes of alcohol administration: (1) oral consumption, or (2) intravenous infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alcohol: Oral administration (Experimental): Participants in this arm will consume a measured dose of alcohol orally, with the goal of achieving a target peak breath alcohol concentration of .065% within 20 minutes.
  Interventions: Drug: Alcohol: Oral administration
- Alcohol: Intravenous administration (Experimental): Participants in this arm will be infused intravenously with a dose of alcohol sufficient to raise their breath alcohol concentration to .065% within 20 minutes.
  Interventions: Drug: Alcohol: Intravenous administration

INTERVENTIONS:
Drug: Alcohol: Oral administration — Patients who plan to undergo bariatric surgery will consume a controlled dose of alcohol orally.
  Arms: Alcohol: Oral administration
Drug: Alcohol: Intravenous administration — Patients who plan to undergo bariatric surgery will be infused with alcohol intravenously.
  Arms: Alcohol: Intravenous administration

SUMMARY:
The study will involve administration of alcohol in a controlled laboratory setting to individuals who are scheduled for Roux-en-Y gastric bypass surgery, and then asking them to return for another laboratory session 3 months following their surgery. A small number will be asked to return again 9 months following their surgery.

The primary objective for this research is to collect pilot data on the effects of metabolic surgery (MS), also known as bariatric surgery, on the metabolism of alcohol. These data will be used as preliminary evidence in support of a subsequent application for funding, to be submitted to the National Institutes of Health.

A secondary objective for this research is to determine the extent to which MS changes reactivity to alcohol-related cues. Heightened reactivity (e.g., attention bias; craving) to alcohol-related cues is known to signify increased risk for heavy drinking and AUD. No research to date has examined whether the increased sensitivity to alcohol that occurs as a result of MS changes cue-reactivity responses, which in theory reflect an individual's history of learning to associate alcohol consumption with its subjective effects.

An exploratory objective is to compare metabolism of alcohol administered orally versus intravenously. IV infusion of alcohol bypasses so-called "first pass metabolism" of alcohol after absorption by the gastrointestinal tract. Thus, compared to oral ingestion, infusion can achieve the same blood alcohol concentration (BAC) with substantially less total alcohol dosage. Following the hypothesis, this should mean that, compared to oral ingestion, infusion will be associated with less production of liver fat, while also mimicking in pre-surgery patients what the investigators observe with oral ingestion following surgery. This comparison will permit better specification of when (during metabolism) and how alcohol is converted to liver fat, and will allow the investigators to separate effects of initial sensitivity to alcohol (a person's subjective response to the initial introduction of alcohol into the body) from effects associated with tolerance (i.e., the body's attempts to re-establish homeostasis after alcohol is introduced).

ELIGIBILITY:
Inclusion Criteria:

* Obese, with body weight less than 450 lbs
* non-smoking female volunteers of any race
* age 30-55 years
* drink alcohol in moderation and meet all of the BSC's indications and criteria for RYGB surgery. NIH/NIAAA criteria specify an average of between 3 and 7 standard drinks per week as moderate alcohol drinking (for women). In addition, included participants must fall within the upper or lower tercile of scores on the ASQ for a bariatric population, as determined by the investigator's previous studies with this population.9,10,19

Exclusion Criteria:

* their AUDIT scores (16 or above) indicate the possibility of a current or prior alcohol use disorder.
* they report typically drinking less than once per month and consuming less than 3-4 drinks per occasion.
* they are taking prescribed psychoactive medications, other than selective serotonin reuptake inhibitors (SSRIs) for anxiety/depression.
* they are taking medications that might interfere with alcohol metabolism (e.g., anti-histamine h2 receptor antagonists [mainly, antacids used to treat GERD and gastro-intestinal ulcers], certain antibiotics such as erythromycin, or other drugs influencing hepatic cytochrome P450 2E1; see medicine.iupui.edu/clinpharm/ddis/table.aspx).
* their medical records indicate current anemia.
* their FTND scores indicate moderate or greater nicotine dependence (4 or above).
* they report they are trying to become pregnant, or produce a positive urine screen for pregnancy at the lab session.
* their body weight is > 450 lbs.
* they have participated in any other research study or medical procedure involving ionizing radiation exposure greater than a chest X-ray in the past 12 months.
* they live more than 60 miles from the CRC.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Subjective Effects of Alcohol Scale | Multiple intervals following alcohol administration, up to 4 hours post-exposure
  Participants' self-reported feelings of stimulation, sedation, and intoxication following exposure to a controlled dose of alcohol in the lab will be assessed using the Subjective Effects of Alcohol Scale (Morean, Corbin, & Treat, 2013). Possible score values range from 0 to 140, where a score of 0 indicates the absence of any subjective feelings related to consumed alcohol. This scale and its psychometric properties were first described in the following publication:
  Morean ME, Corbin WR, Treat TA. The Subjective Effects of Alcohol Scale: development and psychometric evaluation of a novel assessment tool for measuring subjective response to alcohol. Psychol Assess. 2013;25(3):780-795. doi:10.1037/a0032542
Alcohol Urge Questionnaire | Assessed prior to acute alcohol exposure, approximately 10 minutes
  Cue-induced craving for alcohol will be assessed using a beverage presentation procedure. Participants complete a self-report measure of craving, the Alcohol Urge Questionnaire. Participants then are presented with a glass containing an alcoholic beverage and are instructed to pick it up and sniff it 5 times over a 3-min period. Then the AUQ is completed again. Change in AUQ score from baseline to the post-alcohol assessment provides a cue-induced craving score. Scores at each assessment can range from 0 to 48, where 0 indicates the total lack of any craving for alcohol.
  Bohn, M. J., Krahn, D. D., & Staehler, B. A. (1995). Development and initial validation of a measure of drinking urges in abstinent alcoholics. Alcoholism: Clinical and Experimental Research,19(3), 600-606.
Alcohol Sensitivity Questionnaire | Pre-surgery and 3 months after surgery
  Individual differences in self-reported sensitivity to alcohol's effects will be assessed using the Alcohol Sensitivity Questionnaire. This measure contains 15 items, each describing an effect people typically experience when drinking alcohol (e.g., feeling more talkative). For each item, participants indicate (1) whether they have ever experienced the effect in question from drinking alcohol, and (2) if so, the number of standard drinks they typically require in order to experience that effect.
  Fleming, K. A., Bartholow, B. D., Hilgard, J., McCarthy, D. M., O'Neill, S. E., Steinley, D., & Sher, K. J. (2016). The Alcohol Sensitivity Questionnaire: Evidence for construct validity. Alcoholism: Clinical and Experimental Research, 40, 880-888.
Reactivity to alcohol cues: motivational approach bias | Assessed prior to acute alcohol exposure, approximately 10 minutes
  The tendency to approach alcohol-related cues will be assessed using a laboratory task known as the Alcohol Approach-Avoidance Task. In this task, images of alcoholic beverages, nonalcoholic beverages, and non-consumable liquids (e.g., motor oil) are presented on a computer monitor one at a time. Participants are instructed to push or pull on a computer joystick in response to each image, depending on whether it appears to be tilted 3 degrees to the right vs. the left. Each type of image is presented in both orientations multiple times. Approach bias is defined for each image type as the difference in response time for images shown in the 'pull' minus the 'push' condition.
  Wiers, R.W., Rinck, M., Kordts, R., Houben, K., Strack, F. (2010). Re-training automatic action-tendencies to approach alcohol in hazardous drinkers. Addiction, 105, 279-287.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Bartholow, Ph.D., Principal Investigator — University of Missouri-Columbia; Elizabeth J Parks, Ph.D., Principal Investigator — University of Missouri-Columbia; Andrew Wheeler, M.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No